CLINICAL TRIAL: NCT05730517
Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen on Dermis Density and Other Skin Parameters: Double Blind, Placebo-controlled, Randomised Three-way Study Comparing the Efficacy of Two Test Products
Brief Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen on Dermis Density and Other Skin Parameters
Acronym: TO-COSKIN-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Tosla d.o.o. (Industry); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST TO-COSKIN-2 01-2023
Record Dates: First submitted 2023-01-31; First posted 2023-02-16 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Dermis Density; Wrinkles; Skin Hydration; Dermis Thickness; Skin Texture; Skin Elasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (CP5HA Group) (Active Comparator): Participants will receive investigational product 1 containing collagen (5 g/ 15 mL), hyaluronic acid (30 mg/ 15 mL) and vitamin C (80 mg/ 15 mL).
  Interventions: Dietary Supplement: CP5HA
- Placebo group (Placebo Comparator): Placebo group participants will receive placebo syrup without active ingredients. (daily dose 15 mL: collagen: 0 mg, HA: 0 mg, vitamin C: 0 mg); continous administration of placebo product for 12 weeks.
  Interventions: Dietary Supplement: Placebo syrup
- Test group 2 (CP5 Group) (Active Comparator): Participants will receive investigational product 2 containing collagen (5 g/ 15 mL) and vitamin C (80 mg/ 15 mL).
  Interventions: Dietary Supplement: CP5

INTERVENTIONS:
Dietary Supplement: CP5HA — Test group 1 will receive investigational product 1 containing collagen (5 g/ 15 mL), hyaluronic acid (30 mg/ 15 mL) and vitamin C (80 mg/ 15 mL); continuous administration of investigational product for 16 weeks.
  Arms: Test group 1 (CP5HA Group)
Dietary Supplement: Placebo syrup — Placebo group will receive placebo syrup without active ingredients. (daily dose 25 mL: collagen: 0 mg, MSM: 0 mg, vitamin C: 0 mg; continous administration of placebo product for 16 weeks.
  Arms: Placebo group
Dietary Supplement: CP5 — Test group 2 will receive investigational product 2 containing collagen (5 g/ 15 mL) and vitamin C (80 mg/ 25 mL); continuous administration of investigational product for 16 weeks.
  Arms: Test group 2 (CP5 Group)

SUMMARY:
The aim of the randomized, double-blind, placebo-controlled, one-period effectiveness study is to compare the effects of multiple-dose 16 weeks daily dietary supplementation with 5 g collagen alone or 5 g of collagen in combination with hyaluronic acid on skin in healthy human subjects in comparison to placebo product. The main objective is to show that test products have beneficial effects on dermis density, and also on other skin parameters and to investigate differences in the effects among test products.

DETAILED DESCRIPTION:
Single centre, randomized, double-blind, placebo-controlled, one-period effectiveness study will include 84 subjects. Subjects will be divided in three groups, 28 in each. Test group 1 (TG1) will receive investigational product 1 (CP5HA, daily dose 15 mL: collagen 5 g, hyaluronic acid (HA): 30 mg, vitamin C: 80 mg), test group 2 (TG2) will receive investigational product 2 (CP5, daily dose 15 mL: collagen 5 g, vitamin C: 80 mg) and the placebo group (PG) will receive placebo product without those active ingredients (15 mL: 0 g collagen, 0 g HA, 0 g vitamin C). Participants will test continuous administration of placebo or investigational products for 16 weeks in order to demonstrate and assess multiple-dose effects.

ELIGIBILITY:
Inclusion criteria:

* Caucasian female volunteers aged between 40 and 65 years at the time of the signature of Informed consent form (ICF),
* Signed Informed consent form (ICF),
* Fitzpatrick skin phototypes I-IV,
* Signs of skin aging,
* In good general health condition,
* Body mass index (BMI) < 35
* Willingness to avoid a consumption of any food supplements containing hyaluronic acid, methylsulfonylmethane (MSM), antioxidants, collagen and other protein-based food supplements during the study,
* Willingness to follow all study procedures and keeping a diary during the study (to follow their compliance and palatability).
* Willingness to maintain their living habits and to not begin or change any estrogen or progesterone therapies,
* Willingness to avoid shaving/depilation of their arms during the study,
* Willingness not to change cosmetic treatment routine during the study,
* Willingness to avoid rejuvenation treatments during the study.

Exclusion criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products,
* Changes in dietary habits and dietary supplementation in the last three months prior to inclusion,
* Regular use of food supplements containing MSM, antioxidants, collagen or other protein-based food supplements in the last three months prior to inclusion,
* Veganism,
* Changes in cosmetic facial and body care routine in the last month prior to inclusion,
* Diagnosed and uncontrolled/unregulated disease,
* Any clinically significant history of serious metabolic disease, digestive tract disease, liver disease, kidney disease, hematological disease,
* Intake of drugs with any impact on skin reactions (e.g., glucocorticoids, antihistamines, and immunomodulators),
* Any clinically significant acute or chronic skin diseases,
* Skin pigmentation disorders on measuring sites,
* Anticipated sunbathing or solarium visits before or during the study,
* Invasive rejuvenation treatments (e.g. needle rollers, needle mesotherapy, deep/medium-deep chemical peels, abrasive laser treatments etc.) in the last 4 months prior to study entry,
* Non-invasive rejuvenation treatments (e.g. radiofrequency, electrotherapy, ultrasound, intense pulsed light therapy (IPL), non-abrasive laser treatments) in the last month prior to study entry,
* Shaving/depilation of the arms in the last 14 days before inclusion,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 87 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change of dermis density from baseline in all test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Significant change of dermis density from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation with study product is expected. Dermis density will be assessed through ultrasonographic dermis intensity measurement. Differences in change of dermis density between test groups under primary objective conditions will also be evaluated.

SECONDARY OUTCOMES:
Change of wrinkle volume from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of investigational product on periorbital wrinkles after 16 weeks of dietary supplementation will be done using topography measurements. Differences between test groups will also be evaluated.
Change of skin texture from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  For assessments of skin texture topography roughness measurements (Ra, Rq) will be performed. Significant changes from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation is expected. Differences between test groups will also be evaluated.
Change of skin hydration from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational product on skin hydration after 16 weeks of dietary supplementation. Skin hydration measurements will be performed using conductance principle. Differences between test groups will also be evaluated.
Change of dermis thickness from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Significant change of dermis thickness from baseline in test group, in comparison to placebo group after 16 weeks of dietary supplementation with study product is expected. Dermis density will be assessed using ultrasonography. Differences between test groups will also be evaluated.
Change of skin elasticity from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Significant change of skin elasticity from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation with study products is expected. Skin elasticity will be assessed using viscoleasticity measurement (Units of Measure: MPa). Differences between test groups will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — Head of Reasearch Group
Locations (1):
- VIST - Faculty of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No